CLINICAL TRIAL: NCT01385878
Title: Intraoperative Performance & Postoperative Outcomes Following Phacoemulsification With 1.8 & 2.2mm Incision: Randomized Clinical Trial
Brief Title: Outcomes Following Phacoemulsification With 1.8 & 2.2mm Incision: Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Dr. Abhay R. Vasavada, Director, Iladevi Cataract & IOL Research Centre, Iladevi Cataract & IOL Research Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICIRC-1.8 VS 2.2
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Cataract
Keywords: Microcoaxial phacoemulsification, 1.8mm, 2.2mm
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phacoemulsification with 1.8mm incision (Active Comparator): Microcoaxial phacoemulsification was performed using a 1.8mm clear corneal incision
  Interventions: Procedure: Microcoaxial Phacoemulsification
- Phacoemulsification with 2.2mm incisi (Active Comparator): Microcoaxial phacoemulsificaiton will be performed through 2.2mm incision
  Interventions: Procedure: Microcoaxial Phacoemulsification

INTERVENTIONS:
Procedure: Microcoaxial Phacoemulsification — Phacoemulsification through small clear corneal incision
Procedure: Microcoaxial Phacoemulsification — Phacoemulsification through clear corneal incision
Procedure: Microcoaxial Phacoemulsification — Microcoaxial Phacoemulsification through 1.8mm incision
Procedure: Microcoaxial Phacoemulsification — Microcoaxial phacoemulsification through 2.2mm incision
  Arms: Phacoemulsification with 2.2mm incisi

SUMMARY:
Cataract surgical techniques have significantly changed in recent years with the widespread adoption of smaller and smaller clear corneal incisions for phacoemulsification. Microincision surgery has many advantages, including reduced surgically induced astigmatism, faster visual recovery, and reduced intra and postoperative inflammation. Curently, microcoaxial phacoemulsification is being performed through 1.8 as well as 2.2 mm incisions. However, there is still a debate as to which is the best absolute incision size for microcoaxial cataract surgery.

The aim of this study is to evaluate incision stability following microcoaxial phacoemulsification performed through 1.8 and 2.2 mm systems, as well as compare intraoperative performance and postoperative outcomes following microcoaxial phacoemulsification performed through these two incision sizes.

DETAILED DESCRIPTION:
Cataract surgical techniques have significantly changed in recent years with the widespread adoption of smaller and smaller clear corneal incisions for phacoemulsification. Microincision surgery has many advantages, including reduced surgically induced astigmatism, faster visual recovery, and reduced intra and postoperative inflammation. In the recent times, microcoaxial phacoemulsification has gained popularity. The main advantage of this newer technique is that it uses the same methods as the conventional method but with smaller incisions. Curently, microcoaxial phacoemulsification is being performed through 1.8 as well as 2.2 mm incisions. However, there is still a debate as to which is the best absolute incision size for microcoaxial cataract surgery.

The aim of this study is to evaluate incision stability following microcoaxial phacoemulsification performed through 1.8 and 2.2 mm systems, as well as compare intraoperative performance and postoperative outcomes following microcoaxial phacoemulsification performed through these two incision sizes.

ELIGIBILITY:
Inclusion Criteria: Uncomplicated age related cataracts, NO grade II III, IV (LOCS III classification)

-

Exclusion Criteria:

* Ocular comorbidity, glaucoma, uveitis, shallow anterior chamber, maximal pupillary dilatation <6mm, high myopia (axial length > 25mm), previous ocular trauma or surgery, pseudoexfoliation, traumatic cataract, subluxated cataract

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Ingress of Trypan blue from the Ocular Surface into the Anterior Chamber | Immediately at the end of surgery
  At end of surgery, stromal hydration of all incisions will be performed.0.0125% trypan blue will be instilled on the conjunctival surface.After 2 minutes, the surface will be irrigated with balanced salt solution. 0.1ml aqeous aspirate will be obtained from the anterior chamber.Concentration of trypan blue in the aspirate will be ascertained by UV visible spectrophotometry. Log dilutions of concentration of trypan blue will be used for statistical analysis

SECONDARY OUTCOMES:
Surgically Induced Astigmatism | At baseline and 3 months postoperatively
Corneal Endothelial Cell Loss | Baseline and 3 months postoperatively
Change in Central Corneal Thickness | Baseline and 1 week
Anterior Chamber Inflammation | Baseline and 1 week
Anterior Chamber Inflammation | Baseline and 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Abhay R Vasavada, MS, FRCS, Principal Investigator — Iladevi Cataract and IOL Research Center
Locations (1):
- Iladevi Cataract & IOL Research Centre, Ahmedabad, Gujarat, India

REFERENCES:
- [Background] Lee KM, Kwon HG, Joo CK. Microcoaxial cataract surgery outcomes: comparison of 1.8 mm system and 2.2 mm system. J Cataract Refract Surg. 2009 May;35(5):874-80. doi: 10.1016/j.jcrs.2008.12.031. PMID 19393887